CLINICAL TRIAL: NCT05606419
Title: The Crohn's Disease Exclusion Diet With Early Dairy Introduction vs Partial Enteral Nutrition (CD-EDEN) in Adult Patients With Crohn's Disease
Brief Title: The Crohn's Disease Exclusion Diet With Early Dairy Introduction vs Partial Enteral Nutrition for Crohn's Disease
Acronym: CD-EDEN
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was suspended on September 24 because of funding constraints. At that point, approximately 50 % of the planned participants had enrolled. All data collected to date will be analyzed.
Sponsor: Evangelismos Hospital (Other)
Collaborators: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Dimitrios Karayiannis, Chief Dietitian-Nutritionist, Evangelismos Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 605/16-12-2021
Record Dates: First submitted 2022-10-24; First posted 2022-11-04 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease
Keywords: Inflammatory Bowel Diseases; Diet therapy; Crohn's Disease; Enteral Nutrition; Partial Enteral Nutrition; Gastrointestinal Diseases
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: Patients with mildly active disease will follow either the CDED diet protocol (CDED + PEN) or the CDED diet with dairy products included, for up to12 weeks. All participants will attend study visits at the beginning, in the middle and at end of the trials, at which points questionnaires will be completed and samples will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDED + PEN (Experimental): Crohn's Disease Exclusion Diet (CDED)+Partial Enteral Nutrition (PEN): Patients will follow the first phase diet (CDED+50%PEN) for 6 weeks and will continue with CDED phase 2 + 25%PEN for another 6 weeks. Total duration: 12 weeks.
  Interventions: Dietary Supplement: CDED+PEN
- CDED + Dairy (Active Comparator): Crohn's Disease Exclusion Diet (CDED) + dairy products: Patients will follow the first phase diet CDED + 50% of their energy requirements covered by dairy products for 6 week and then will continue with the CDED phase 2 diet + 25% dairy products.
  Interventions: Dietary Supplement: CDED+dairy

INTERVENTIONS:
Dietary Supplement: CDED+PEN — Dietary intervention (Liquid food replacement intervention and specific exclusion diet). Focus on 24 hour diet recalls to asses adherence.
  Arms: CDED + PEN
Dietary Supplement: CDED+dairy — Dietary intervention (Specific exclusion diet plus early dairy introduction). Focus on 24 hour diet recalls to asses adherence.
  Arms: CDED + Dairy

SUMMARY:
This study aims to evaluate a novel diet for adult Crohn's disease patients (The Crohn's Disease Exclusion Diet - CDED). Some of the patients in this study will receive the CDED combined with partial enteral nutrition (PEN), while the other group will receive the CDED with early introduction of dairy products, that were eliminated from the initial CDED protocol.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic relapsing inflammatory bowel disease that has a significant impact on patients' quality of life and is of increased incidence worldwide. The disease aetiology is complex and not fully understood. Accumulated data indicate that environmental factors, including diet, might play a key role in the pathogenesis and inflammation, through mechanisms involving gut dysbiosis, in genetically susceptible people. Epidemiological data suggest that a Mediterranean dietary pattern is associated with decreased risk for CD, whereas a Western diet, rich in animal fat, processed foods and food additives, seems to be linked with an increased disease risk.

Exclusive Enteral Nutrition (EEN) is the only well-established dietary therapy in CD and is used as the first line therapy for the induction of remission in mild to moderate pediatric CD. Evidence according to EEN efficacy in adults is not consistent, which could partly be explained by the compliance difficulty. It is of interest, that feacal inflammation increases rapidly after food re-introduction following EEN in children. Partial enteral nutrition (PEN) has been shown to be beneficial in maintaining remission, but poor compliance due to low formula palatability and patients' fatigue remains an important barrier in the clinical practice. Moreover, PEN is inferior to EEN in inducing remission. Crohn's Disease Exclusion Diet (CDED), which eliminates specific dietary components hypothesized to induce dysbiosis, appears to be effective in inducing and maintaining remission both in pediatric and adult populations. In parallel, patients express a strong interest in ways to manage their disease through diet, so the establishment of a palatable and as flexible as possible dietary pattern, not merely for inducing remission, but also as a feasible maintenance strategy is one of the main priorities in CD research at present.

Therefore, the aim of this study is to explore the effectiveness of the CDED and PEN in both inducing and maintaining remission of CD in adults. The investigators also wish to challenge patients with an early exposure to dairy products, to assess tolerability, prospecting for the development of a more flexible dietary approach based on the CDED principles. The investigators aim to assess the intervention effect on CD activity, based on routinely used clinical indices, blood and faecal inflammatory biomarkers (CRP, FC), health-related quality of life, nutritional status and dietary intake, in patients with mildly active CD.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have an established diagnosis of CD
* Participants must have clinically active disease defined as HBI ≥ 5
* Participants must have confirmed inflammation at screening as CRP > 5 mg/L, FC >100 mg/g, or presence of inflammation on endoscopy in the 3 months before screening based on retrospective review of procedure reports by the local investigator and the clinician's assessment
* Individuals able to give informed consent and willingness to participate

Exclusion Criteria:

* Age < 18 years old
* Previous extensive bowel resection
* Reported pregnancy or lactation
* Current stoma
* Current abscess
* Clinically significant stricture
* Introduction of or change in dose of drug therapy within the past 8 weeks
* Comorbidities including diabetes or coeliac disease, or other concomitant serious comorbidity e.g. significant psychiatric, hepatic, renal, endocrine, respiratory, neurological, cardiovascular, neoplastic or other autoimmune disease
* Food allergies or intolerances, which do not permit participation in the study
* Any proven current infection such as positive stool cultures or positive tests for parasites or C. difficile. Stool tests are mandatory only if diarrhea is present.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Clinical response - Change in Harvey Bradshaw Index (HBI) | Baseline, 6 weeks, 12 weeks
  Higher HBI scores indicate worse outcomes. Clinical response is defined as baseline HBI score decrease of ≥ 3, and clinical remission is defined as score <5

SECONDARY OUTCOMES:
Faecal calprotectin | Baseline, 6 weeks, 12 weeks
  Change in faecal calprotectin level
Change in serum CRP | Baseline, 6 weeks, 12 weeks
  Abnormal/higher values indicate worse outcomes.
Change in serum Albumin | Baseline, 6 weeks, 12 weeks
  Abnormal values indicate worse outcomes
Bowel symptoms improvement | Baseline, 6 weeks, 12 weeks
  Percent of patients who reported improvement in bowel symptoms, assessed by the validated IBDQ (bowel symptoms domain: 10 questions)
Health Related Quality of Life (HR-QoL) | Baseline, 6 weeks, 12 weeks
  HR-QoL defined by the self-administered Inflammatory Bowel Disease questionnaire (IBDQ) score. Higher IBDQ scores indicate better outcomes. Clinical response defined as increase ≥16 points.
Patient's tolerance to the diet | Baseline, 6 weeks, 12 weeks
  Intolerance: patient's refusal to continue diet (based on reporting and the 24 hour recalls); Adherence will be assessed based on the modified Medication Adherence Report Scale (MARS) questionnaire; The modified MARS questionnaire rates how closely patients adhere to the diet. A score of 1-5 indicates that the patient is not adherent; a score of 6-9 indicates that the patient is adherent.
Weight (kg) | Baseline, 6 weeks, 12 weeks
  Comparison of body weight between the groups.
Body mass index (BMI) (kg/m^2) | Baseline, 6 weeks, 12 weeks
  Comparison of Body Mass Index (BMI) (kg/m2) between the groups.
Waist circumference (WC) (cm) | Baseline, 6 weeks, 12 weeks
  Comparison of WC between groups.
Handgrip strength (kg) | Baseline, 6 weeks, 12 weeks
  Handgrip strength measured with handgrip strength dynamometer
Neck circumference (cm) | Baseline, 6 weeks, 12 weeks
  Comparison of neck circumference measured with tape measure between the groups
Mid arm circumference (MAC) (cm) | Baseline, 6 weeks, 12 weeks
  Measured with tape measure to assess Mid-arm muscle circumference (MAMC) (for estimating FFM, when BIA is not feasible)
Triceps Skinfold (TSF) (mm) | Baseline, 6 weeks, 12 weeks
  Measured with a skinfold caliper to assess Mid-arm muscle circumference (MAMC) for estimating FFM, when BIA in not feasible)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Karayiannis, Dr., Principal Investigator — Evangelismos General Hospital of Athens; Kalliopi Anna Poulia, Dr., Study Director — Agricultural University of Athens; Gerasimos Mantzaris, Dr., Study Chair — Evangelismos General Hospital of Athens; Nikos Viazis, Dr., Study Chair — Evangelismos General Hospital of Athens
Locations (1):
- Evangelismos General Hospital of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gkikas K, Gerasimidis K, Milling S, Ijaz UZ, Hansen R, Russell RK. Dietary Strategies for Maintenance of Clinical Remission in Inflammatory Bowel Diseases: Are We There Yet? Nutrients. 2020 Jul 7;12(7):2018. doi: 10.3390/nu12072018. PMID 32645980
- [Background] Levine A, Sigall Boneh R, Wine E. Evolving role of diet in the pathogenesis and treatment of inflammatory bowel diseases. Gut. 2018 Sep;67(9):1726-1738. doi: 10.1136/gutjnl-2017-315866. Epub 2018 May 18. PMID 29777041
- [Background] Bischoff SC, Escher J, Hebuterne X, Klek S, Krznaric Z, Schneider S, Shamir R, Stardelova K, Wierdsma N, Wiskin AE, Forbes A. ESPEN practical guideline: Clinical Nutrition in inflammatory bowel disease. Clin Nutr. 2020 Mar;39(3):632-653. doi: 10.1016/j.clnu.2019.11.002. Epub 2020 Jan 13. PMID 32029281
- [Background] Wall CL, Day AS, Gearry RB. Use of exclusive enteral nutrition in adults with Crohn's disease: a review. World J Gastroenterol. 2013 Nov 21;19(43):7652-60. doi: 10.3748/wjg.v19.i43.7652. PMID 24282355
- [Background] Logan M, Clark CM, Ijaz UZ, Gervais L, Duncan H, Garrick V, Curtis L, Buchanan E, Cardigan T, Armstrong L, Delahunty C, Flynn DM, Barclay AR, Tayler R, McDonald E, Milling S, Hansen RK, Gerasimidis K, Russell RK. The reduction of faecal calprotectin during exclusive enteral nutrition is lost rapidly after food re-introduction. Aliment Pharmacol Ther. 2019 Sep;50(6):664-674. doi: 10.1111/apt.15425. Epub 2019 Jul 25. PMID 31342536
- [Background] Yang H, Feng R, Li T, Xu S, Hao X, Qiu Y, Chen M. Systematic review with meta-analysis of partial enteral nutrition for the maintenance of remission in Crohn's disease. Nutr Res. 2020 Sep;81:7-18. doi: 10.1016/j.nutres.2020.06.006. Epub 2020 Jun 9. PMID 32798791
- [Background] Levine A, Wine E, Assa A, Sigall Boneh R, Shaoul R, Kori M, Cohen S, Peleg S, Shamaly H, On A, Millman P, Abramas L, Ziv-Baran T, Grant S, Abitbol G, Dunn KA, Bielawski JP, Van Limbergen J. Crohn's Disease Exclusion Diet Plus Partial Enteral Nutrition Induces Sustained Remission in a Randomized Controlled Trial. Gastroenterology. 2019 Aug;157(2):440-450.e8. doi: 10.1053/j.gastro.2019.04.021. Epub 2019 Jun 4. PMID 31170412
- [Background] Yanai H, Levine A, Hirsch A, Boneh RS, Kopylov U, Eran HB, Cohen NA, Ron Y, Goren I, Leibovitzh H, Wardi J, Zittan E, Ziv-Baran T, Abramas L, Fliss-Isakov N, Raykhel B, Gik TP, Dotan I, Maharshak N. The Crohn's disease exclusion diet for induction and maintenance of remission in adults with mild-to-moderate Crohn's disease (CDED-AD): an open-label, pilot, randomised trial. Lancet Gastroenterol Hepatol. 2022 Jan;7(1):49-59. doi: 10.1016/S2468-1253(21)00299-5. Epub 2021 Nov 2. PMID 34739863

DOCUMENTS (1):
  • Informed Consent Form (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT05606419/ICF_001.pdf